CLINICAL TRIAL: NCT05871307
Title: Neoadjuvant vs. Intraoperative vs. Adjuvant Resection Cavity Radiotherapy of Brain Metastases - A Prospective Randomized Explorative Phase II Trial
Brief Title: Neoadjuvant vs. Intraoperative vs. Adjuvant Resection Cavity Radiotherapy of Brain Metastases
Acronym: Radcav
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Department Director, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADOnk-Radcav
Record Dates: First submitted 2022-11-02; First posted 2023-05-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Brain Metastases; Radiotherapy
Keywords: Brain Metastases; Radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Arm A (Preoperativ SRS) (Experimental): Preoperative stereotatic radiosurgery following resection of brain metastases after 1-7 days
  Interventions: Radiation: Preoperative Radiotherapy
- Experimental Arm B (Intraoperativ SRS) (Experimental): Intraoperative stereotactic radiotherapy after resection of brain metastases
  Interventions: Radiation: Intraoperative Radiation
- Standard Treatment Arm C (Posoperativ SRS) (Active Comparator): Resection of brain metastases following stereotactic radiotherapy after 2-6 weeks
  Interventions: Radiation: Postoperative Radiotherapy

INTERVENTIONS:
Radiation: Preoperative Radiotherapy — Resection of brain mestases following
  Arms: Experimental Arm A (Preoperativ SRS)
Radiation: Intraoperative Radiation — While Resection
  Arms: Experimental Arm B (Intraoperativ SRS)
Radiation: Postoperative Radiotherapy — After resection
  Arms: Standard Treatment Arm C (Posoperativ SRS)

SUMMARY:
Patients suffering from malignancies in advanced stages often develop brain metastases, which limit both the life span and the quality of life.

Combining surgery and radiotherapy for resectable brain metastases is standard of care but there is a lot of controversy on which kind of radiotherapy is best suitable. Recently, first volumetric in-silico analyses point to theoretical advantages of neoadjuvant stereotactic radiotherapy of brain metastases. Special about this trial is the direct comparison between the three currently discussed radiotherapy options for resectable brain metastases: Neoadjuvant stereotactic radiotherapy, intraoperative radiotherapy and adjuvant stereotactic radiotherapy.

DETAILED DESCRIPTION:
This trial approach allows for detailed comparison of resected tissue samples, cerebrospinal fluid and blood of all patient groups. So, the investigators will investigate biomaterial of recently irradiated (neoadjuvant and intraoperative arms) and non-irradiated (adjuvant arm) tissue. All this prompts the main issues of the explorative randomized controlled phase 2 RADCAV trial: Is there a difference between neoadjuvant stereotactic radiotherapy vs. intraoperative radiotherapy vs. adjuvant stereotactic radiotherapy regarding the factors immune profiling, dosimetry, efficacy and toxicity. It can be hypothesized that the resected tissue differs between recently irradiated and non-irradiated brain metastases, for example regarding different histopathologic and molecular pathologic markers including immune environment, markers for cell death and markers for tumor invasion. Are there histopathologic and molecular pathologic markers of tumor cell response and prognosis so the investigators can better understand the effects of irradiation on metastatic brain tissue? And are there relevant differences in dosimetry that put patients at different risks for efficacy and toxicity?

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid malignancy

  * Metastatic brain disease (1-10 brain metastases), with at least one brain metastasis in a non-eloquent location (i.e. motor or speech) planned for resection
  * Maximum size of the brain metastasis <5cm
  * Eligibility of patients for both stereotactic radiotherapy and resection
  * Time interval from resection to adjuvant stereotactic radiosurgery of 2-6 weeks
  * Time interval from neoadjuvant stereotactic radiosurgery to resection of 1-7 days
  * Possibility to postpone resection for neoadjuvant stereotactic radiosurgery, if applicable
  * Karnofsky performance scores >= 70 or Eastern Cooperative Oncology Group (ECOG) >= 2 at enrollment
  * Age ≥ 18 years of age
  * For women with childbearing potential, (and men) adequate contraception.
  * Ability of subject to understand character and individual consequences of the clinical trial
  * Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

Necessity of immediate surgical resection due to life threatening symptoms

* brain metastasis directly located (≤10mm) next to the optic system or brain stem
* Refusal of the patients to take part in the study
* Small-cell lung cancer (SCLC) or hematologic malignancy as primary malignant illness
* Leptomeningeal disease suspected RadCav Trial Protocol Version 1.1, 01.07.2022 18
* Previous radiotherapy of the brain
* Contraindication for contrast-enhanced MRI
* Pregnant or lactating women
* Participation in another competing clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of treatment response | through study completion, an avarage of 60 month
  number of patients without progresion according to RANO-BM
local tumor control | through study completion, an avarage of 60 month
  events of tumor progression or recurrence in the area of 1cm surrounding the resection cavity and surrounding the surgical access

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Debus, Prof., Principal Investigator — University Hospital of Heidelberg, Radiation Oncology
Locations (1):
- Department of Radiotherapy, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No